CLINICAL TRIAL: NCT02100553
Title: A Phase 1, Open Label, Two Period, Fixed Sequence, Parallel Group Study To Estimate The Effects Of Multiple Dose Administration Of Itraconazole On The Single Dose Pharmacokinetics Of Conjugated Estrogens/Bazedoxifene In Non Obese (Bmi <30 Kg/m2) And Obese (Bmi ≥30 Kg/m2) Postmenopausal Women
Brief Title: Study Evaluating Effects of Multiple-Dose Administration of Itraconazole on the Single Dose Pharmacokinetics of Conjugated Estrogens/Bazedoxifene in Non-Obese and Obese Postmenopausal Women
Acronym: CE/BZA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B2311065
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Postmenopausal Women; Obese; Non-obese; Drug Interaction with Itraconazole; Pharmacokinetic
MeSH Terms: conditions — Obesity | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Obese (Other): BMI <30 kg/m^2
  Interventions: Drug: CE/BZA; Drug: Itraconazole
- Obese (Other): BMI >= 30 kg/m^2
  Interventions: Drug: CE/BZA; Drug: Itraconazole

INTERVENTIONS:
Drug: CE/BZA — CE 0.45mg/BZA 20mg tablets, single dose
  Other Names: Duavee
  Arms: Non-Obese
Drug: Itraconazole — Two 100 mg capsules, once daily for 7 days
  Other Names: Sporanox
  Arms: Non-Obese
Drug: CE/BZA — CE 0.45mg/BZA 20mg tablets, single dose on Day 5
  Other Names: Duavee
  Arms: Non-Obese
Drug: CE/BZA — CE 0.45mg/BZA 20mg tablets, single dose
  Other Names: Duavee
  Arms: Obese
Drug: Itraconazole — Two 100 mg capsules, once daily for 7 days
  Other Names: Sporanox
  Arms: Obese
Drug: CE/BZA — CE 0.45mg/BZA 20mg tablets, single dose on Day 5
  Other Names: Duavee
  Arms: Obese

SUMMARY:
This study will assess if itraconazole will affect the blood levels of Duavee when they are given together. This study will also assess if a subject's body size affects the blood levels of Duavee.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy postmenopausal women, aged 40-64. Intact Uterus

Exclusion Criteria:

* The use of oral, vaginal, or transdermal estrogen, androgen or progestin-containing medications within 30 days before study drug administration.

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] for BZA, total estrone adjusted for baseline and total equilin. | up to 96 hours
  AUC (0 - inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf).
Maximum Observed Plasma Concentration (Cmax) for BZA, total estrone adjusted for baseline and total equilin. | up to 96 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] for unconjugated estrone, unconjugated estrone adjusted for baseline, total estrone, and unconjugated equilin. | up to 96 hours
  AUC (0 - inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf).
Maximum Observed Plasma Concentration (Cmax) for unconjugated estrone, unconjugated estrone adjusted for baseline, total estrone, and unconjugated equilin. | up to 96 hours
Apparent Oral Clearance (CL/F) for all analytes. | up to 96 hours
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time to Reach Maximum Observed Plasma Concentration (Tmax) for all analytes. | up to 96 hours
Apparent Volume of Distribution (Vz/F) for all analytes. | up to 96 hours
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Terminal Phase Elimination Half-Life (t1/2) for all analytes. | up to 96 hours
  Terminal Phase Elimination Half-Life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - SeaView Research, Inc. (Screening Office), Miami, Florida
  - SeaView Research, Inc., Miami, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2311065&StudyName=Study%20Evaluating%20Effects%20of%20Multiple-Dose%20Administration%20of%20Itraconazole%20on%20the%20Single%20Dose%20Pharmacokinetics%20of%20Conjugated%20Estrogens/Bazedoxifen